CLINICAL TRIAL: NCT02809157
Title: Non-invasive Fractional Flow Reserve CT (FFRCT) Scan for the Study of Coronary Vaso-motion
Brief Title: Non-invasive Fractional Flow Reserve CT (FFRCT)Scan for the Study of Coronary Vaso-motion
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: National Heart Centre Singapore (Other)
Responsible Party: Sponsor
Other Study IDs: 2014/488/c
Record Dates: First submitted 2016-05-31; First posted 2016-06-22 (Estimated); Last update posted 2016-06-22 (Estimated); Status verified 2016-05

CONDITIONS: Coronary Artery Disease
MeSH Terms: conditions — Coronary Artery Disease

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

SUMMARY:
Coronary artery disease (CAD) is a very common cause of heart failure affecting millions of people worldwide, which is caused by build-up of plaque inside arteries of the heart. Build-up of plaque eventually impacts the blood supply to the heart. In medicine, techniques (invasive or non-invasive) such as coronary angiography, intravascular ultrasound, computed tomography, magnetic resonance imaging, positron emission tomography and transthoracic echocardiography can be used to diagnose CAD.

The investigators aim to study Coronary Artery Disease significance with the combination of computed tomography angiography (CTA), and computational fluid dynamics (CFD) methods. CTA is a non-invasive technique to visualize arterial vessels, which uses computer-processed x-rays. Computational Fluid Dynamics employs digital computers and numerical methods to solve complex flow patterns inside arterial vessels. Combining these two methods, the investigators are able to provide detailed blood flow information and mechanical stress distributions on the vessels. This study therefore, aims to propose a non-invasive methodology to assess the significance of CAD.

DETAILED DESCRIPTION:
Cardiovascular disease is the leading cause of death in Singapore, and accounts for 31.9% of all deaths in 2010. Coronary vascular dysfunction has been linked to the development of cardiovascular-related events, such as death, myocardial infarction (MI), stroke and unstable angina. Recently, impaired coronary vaso-motion has been suggested as an independent predictor of poor prognosis, which can predict cardiovascular events in patients with epicardial Coronary Artery Disease . Coronary vaso-motion refers to the change in diameter of a coronary vessel in response to vasoactive agent, which is measured via quantitative coronary angiography (QCA). Better coronary vaso-motion response has been associated with improved survival for both obstructive and non-obstructive CAD.

Another widely used invasive clinical imaging technology to assess CAD is intravascular ultrasound (IVUS), which uses ultrasound technology for imaging the endothelium of vessels. Since detailed histological information of plaques on the endothelium of coronary arteries can be provided by IVUS, it is used as gold standard in evaluating progression or regression of plaque.

Although coronary vaso-motion, FFR and IVUS have been shown to improve clinical outcomes and procedural cost-efficiency in terms of guiding percutaneous interventions, they are invasive procedures. Non-invasive option for the diagnosis of myocardial ischemia is required to relief the patients' pain and medical cost due to the invasive cath. This study aims to fill in the gap. The investigators hypothesize that non-invasive FFRCT can be obtained by combining CT images and CFD methods, which can be used to assess the physiologic significance of CAD.

ELIGIBILITY:
Inclusion Criteria:

1. Aged 21-98.
2. Undergoing coronary angiography, who had received coronary CTA within 2 months before the scheduled coronary angiography.

Exclusion Criteria:

1. Individuals unable to provide informed consent.
2. Non-cardiac illness with life expectancy <2 years.
3. Pregnant or breastfeeding state. Female patients who have a chance of becoming pregnant will receive pregnancy testing to exclude pregnant women from entering the study.
4. Allergy to iodinated contrast.
5. Significant arrhythmia; heart rate ≥ 100 beats/min; systolic blood pressure ≤90 mmHg.
6. Renal dysfunction (Glomerular filtration rate (GFR) <30 mL/min/1.73m2).
7. Contraindication to beta blockers or nitroglycerin.
8. Canadian Cardiovascular Society class IV angina.
9. Significant valvular pathology
10. Previous coronary artery bypass surgery
11. Previous Percutaneous coronary intervention
12. Contraindication to adenosine administration (e.g. asthma, chronic obstructive pulmonary disease, heart rate <50 beats/min)
13. Patients with an acute myocardial infarction or unstable arrhythmias
14. Patients with a left ventricular ejection fraction less than 30%

Ages: 21 Years to 98 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with diagnosed Coronary Artery Disease
Sampling Method: Non-Probability Sample
Enrollment: 10 (Estimated)
Dates: Start 2014-10; Primary Completion 2017-05 (Estimated); Study Completion 2017-05 (Estimated)

PRIMARY OUTCOMES:
Result of combining CT and CFD helps to provide 3D streamlines,pressure and non-invasive FFRCT. | Through study completion (09-May-2017)

CONTACTS AND LOCATIONS:
Overall Officials: A/Prof Tan Ru San, Principal Investigator — National Heart Centre Singapore

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] von Mering GO, Arant CB, Wessel TR, McGorray SP, Bairey Merz CN, Sharaf BL, Smith KM, Olson MB, Johnson BD, Sopko G, Handberg E, Pepine CJ, Kerensky RA; National Heart, Lung, and Blood Institute. Abnormal coronary vasomotion as a prognostic indicator of cardiovascular events in women: results from the National Heart, Lung, and Blood Institute-Sponsored Women's Ischemia Syndrome Evaluation (WISE). Circulation. 2004 Feb 17;109(6):722-5. doi: 10.1161/01.CIR.0000115525.92645.16. PMID 14970106
- [Background] Widlansky ME, Gokce N, Keaney JF Jr, Vita JA. The clinical implications of endothelial dysfunction. J Am Coll Cardiol. 2003 Oct 1;42(7):1149-60. doi: 10.1016/s0735-1097(03)00994-x. PMID 14522472
- [Background] Quyyumi AA. Prognostic value of endothelial function. Am J Cardiol. 2003 Jun 19;91(12A):19H-24H. doi: 10.1016/s0002-9149(03)00430-2. PMID 12818731
- [Background] Sarno G, Bruining N, Onuma Y, Garg S, Brugaletta S, De Winter S, Regar E, Thuesen L, Dudek D, Veldhof S, Dorange C, Garcia-Garcia HM, Ormiston JA, Serruys PW. Morphological and functional evaluation of the bioresorption of the bioresorbable everolimus-eluting vascular scaffold using IVUS, echogenicity and vasomotion testing at two year follow-up: a patient level insight into the ABSORB A clinical trial. Int J Cardiovasc Imaging. 2012 Jan;28(1):51-8. doi: 10.1007/s10554-010-9769-y. Epub 2011 Jan 7. PMID 21213050
- [Background] Halcox JP, Schenke WH, Zalos G, Mincemoyer R, Prasad A, Waclawiw MA, Nour KR, Quyyumi AA. Prognostic value of coronary vascular endothelial dysfunction. Circulation. 2002 Aug 6;106(6):653-8. doi: 10.1161/01.cir.0000025404.78001.d8. PMID 12163423
- [Background] Pijls NH, van Son JA, Kirkeeide RL, De Bruyne B, Gould KL. Experimental basis of determining maximum coronary, myocardial, and collateral blood flow by pressure measurements for assessing functional stenosis severity before and after percutaneous transluminal coronary angioplasty. Circulation. 1993 Apr;87(4):1354-67. doi: 10.1161/01.cir.87.4.1354. PMID 8462157
- [Background] Samady H, Eshtehardi P, McDaniel MC, Suo J, Dhawan SS, Maynard C, Timmins LH, Quyyumi AA, Giddens DP. Coronary artery wall shear stress is associated with progression and transformation of atherosclerotic plaque and arterial remodeling in patients with coronary artery disease. Circulation. 2011 Aug 16;124(7):779-88. doi: 10.1161/CIRCULATIONAHA.111.021824. Epub 2011 Jul 25. PMID 21788584
- See also: Report on Registration of Births and Deaths in 2011 by the Registry of Births and Deaths,Immigration and Checkpoints Authority,Singapore — http://www.myheart.org.sg/article/about-the-heart-and-heart-disease/statistics/singapore/75